CLINICAL TRIAL: NCT01241149
Title: Prospective Evaluation of Symptom Resolution in Acid Versus Non-acid Reflux Disease Following Anti-reflux Surgery.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit a sufficient number of subjects.
Sponsor: United States Naval Medical Center, Portsmouth (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIP# 10.0090
Record Dates: First submitted 2010-11-15; First posted 2010-11-16 (Estimated); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Non-acid Reflux Disease
Keywords: Nissen fundoplication; non-acid reflux disease; anti-reflux surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Normal pH, abnormal Impedance (Active Comparator): After 24hr pH-metry and impedance, those patients with normal pH (i.e. DeMeester score <14.7) but with abnormal impedance scores will be offered anti-reflux surgery
  Interventions: Procedure: anti-reflux surgery
- Abnormal pH (Placebo Comparator): After 24hr pH-metry and impedance, those with abnormal pH scores (i.e. DeMeester score >14.7)will be offered anti-reflux surgery
  Interventions: Procedure: anti-reflux surgery

INTERVENTIONS:
Procedure: anti-reflux surgery — Anti-reflux surgery (Laparoscopic Nissen Fundoplication)

SUMMARY:
Gastroesophageal reflux disease (GERD) is a common ailment affecting a significant portion of the US population. With the advent and increased use of esophageal impedance monitoring, both acid and nonacid reflux disease can be better diagnosed and treated. Patients with severe symptoms or symptoms refractory to medical management may be offered anti-reflux surgery for optimal treatment. Though there are a handful of studies evaluating the efficacy of anti-reflux surgery on those patients with acid or non-acid related reflux disease, the comparison between acid and non-acid reflux disease following surgery is lacking. We propose a prospective study comparing clinical outcomes from those patients with acid versus non-acid reflux disease following anti-reflux surgery with the use of validated and disease specific quality of life surveys.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are offered anti-reflux surgical treatment with elevated DeMeester scores or with low (less than 14.7) DeMeester scores, but with positive impedance scores (positive symptom index associated with reflux episodes).

Exclusion Criteria:

* • Previous major upper gastrointestinal surgery (includes esophagus, stomach, and duodenum) - previous cholecystectomy (gallbladder removal) is not considered a major upper GI surgery

  * Presence of paraesophageal hernia (type II - type IV)
  * Presence of large hiatal hernia >5cm
  * Presence of peptic strictures
  * History of severe esophageal motility disorders such as:

    * achalasia
    * diffuse esophageal spasms
    * scleroderma
    * poorly-controlled diabetes mellitus
    * autonomic or peripheral neuropathy
    * myopathy
  * Pregnancy (As a standard operating procedure, women of child-bearing age will undergo a urine pregnancy test the morning of surgery because anti-reflux surgery is considered an elective case, where pregnancy is a relative contraindication.)
  * BMI greater than 40
  * Undergoes Collis gastroplasty during surgery
  * Conversion to an open procedure
  * Age less than 18 years old

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2014-03-26 (Actual); Study Completion 2014-03-26 (Actual)

PRIMARY OUTCOMES:
Effectiveness of anti-reflux surgery | 1 year
  To prospectively evaluate the effectiveness of anti-reflux surgery, as measured by symptom reduction, in the treatment of nonacid reflux disease compared prospectively with acid reflux disease.

CONTACTS AND LOCATIONS:
Overall Officials: Ellie Mentler, MD, Principal Investigator — United States Naval Medical Center, Portsmouth
Locations (1):
- Naval Medical Center Portsmouth, Portsmouth, Virginia, United States